CLINICAL TRIAL: NCT07315581
Title: Does Age Matter? Outcomes of Pilon Fracture Fixation in Patients Above and Below 40 Years: A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed El-Desouky, Associate Professor of Orthopedic Surgery, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS-62-2021
Record Dates: First submitted 2025-12-11; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pilon Fracture of Tibia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients < 40 years (Active Comparator): Patients in this group had staged ORIF of pilon fracture in younger age
  Interventions: Procedure: staged ORIF of pilon fracture
- Patients 40 years or older (Experimental): Patients in this group had staged ORIF of pilon fracture
  Interventions: Procedure: staged ORIF of pilon fracture

INTERVENTIONS:
Procedure: staged ORIF of pilon fracture — Early application of external fixator followed by open reduction & internal fixation after 10-21 days

SUMMARY:
Pilon fractures are severe intra-articular injuries in the distal tibial plafond that result primarily from high-energy axial compression mechanisms such as road traffic accidents or falls from height [1]. They constitute 1-10% of all tibial fractures and frequently involve significant comminution and compromise of the soft-tissue envelope [1,2]. Successful management requires anatomical reduction of the articular surface, restoration of limb alignment, and careful protection of the soft tissues [3].

Since the first description of open reduction and internal fixation (ORIF) for Pilon fractures by Rüedi and Allgöwer in 1969, surgical protocols have evolved from single-stage fixation to a more conservative two-stage approach to reduce wound complications [4-6]. Despite technical advances, treatment outcomes can vary depending on patient-specific factors such as age, comorbidities, and bone quality [7,8].

Younger patients generally exhibit higher bone density and faster healing potential, while patients above 40 years may experience delayed union, increased risk of infection, and reduced functional recovery due to poorer bone perfusion and degenerative changes [9-11]. However, there is limited comparative data examining the impact of age on the success of ORIF in Pilon fractures.

The current study aims to compare clinical and radiographic outcomes of ORIF in patients below and above 40 years, analyzing differences in union rate, complications, and functional recovery using standardized scoring systems.

ELIGIBILITY:
Inclusion Criteria:

* Closed, fracture
* Complete articular fracture
* Neither 43-C1, 43-C2, or 43-C3 types based on OTA/AO classification

Exclusion Criteria:

* Open fractures
* Pathological fractures
* Acute compartment syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Healing rate | 6 months postoperatively
  Number of cases in which complete healing was achieved

SECONDARY OUTCOMES:
AOFAS | 2 YEARS postoperatively
OMS | 2 YEARS postoperatively
Complications rate | 2 years postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo, Egypt